CLINICAL TRIAL: NCT04133389
Title: Believing People Can Change: An Examination of the Role of Implicit Theory, Attributional Style and Psychological Flexibility in Depression and Wellbeing, & a Randomized Controlled Trial of an Incremental Theory Intervention in Adolescence
Brief Title: Believing People Can Change: A Randomized Controlled Trial of an Incremental Theory Intervention in Adolescence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Margaret Lumley, Associate Professor, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 19-03-019
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Depressive Symptoms; Happiness; Life Satisfaction
Keywords: Growth mindset; Implicit theory; Adolescence; Mental Health; Well-being; students; Secondary Schools; Educational intervention
MeSH Terms: conditions — Depression; Personal Satisfaction; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The current study is a two-wave randomized controlled trial that employs a 2 (group - between participants) by 2 (time - within participants) mixed measures design to assess a brief online implicit theory of personality intervention.
Who Masked: Participant, Investigator
Masking Description: Participants will not be informed that there are different versions of the educational program and thus will be blind to group allocation. Randomization will be fully automated by the online intervention administration system such that researchers will also be blind to group allocation during intervention administration as well as during pre- and post-intervention data collection. Because randomization is automated, neither researchers nor participants will be able to predict randomization assignments. Outcomes will be measured quantitatively thus no assessment of primary outcomes will take place. However, assessors of the manipulation check (which codes for participant engagement in the intervention) will not be masked and thus will be aware of allocation (experimental or control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Growth Mindset of Personality (Experimental): Experimental intervention
  Interventions: Other: Growth mindset of personality educational intervention
- Growth Mindset of Athletic Ability (Placebo Comparator): Control intervention
  Interventions: Other: Growth mindset of athletic ability educational intervention

INTERVENTIONS:
Other: Growth mindset of personality educational intervention — This is a brief online educational intervention that teaches growth mindset of personality. The intervention includes pictures, text, videos, and questions administered through Qualtrics survey software.
  Arms: Growth Mindset of Personality
Other: Growth mindset of athletic ability educational intervention — This is a brief online educational intervention that teaches growth mindset of athletic ability. The intervention includes pictures, text, videos, and questions administered through Qualtrics survey software.
  Arms: Growth Mindset of Athletic Ability

SUMMARY:
This study will test the effectiveness of a brief educational intervention that teaches youth that they can grow and change, known as "growth mindset." Similar growth mindset interventions have improved youths' well-being and academic skills, and reduced risk for depression. In this study, youths' depressive symptoms and well-being will be measured before the intervention and then again 4 months after the intervention to determine if the intervention had a positive impact for youth experiencing transitions (firs and last years of high school).

DETAILED DESCRIPTION:
Adolescents experience many major life transitions during high school, including changes in educational settings, living arrangements, and social and romantic relationships. While these transitions may be experienced as positive new beginnings for some youth, others experience them as stressful and challenging. Further, the developmental period of adolescence is characterized by an increased risk for the development of mental illnesses such as depression. In the context of widely-accepted cognitive models of adolescent depression, adolescents with pre-existing vulnerabilities for depression (e.g., negative self beliefs) may be more prone to experience certain life transitions as especially stressful, and this vulnerability/environment combination is likely to bring about depressive symptomatology for vulnerable youth. Thus, there is a pressing need to better understand factors that not only protect youth from mental illness during transitions, but also factors that promote resilience and well-being. Indeed, high schools are eager to address student mental illness and find better ways of promoting mental health and well-being in schools.

This project employs clinical, cognitive, developmental, and positive psychology theories in an attempt to better understand factors that may be important for adolescent mental illness and mental health during this important time of transition. Specifically, we aim to examine the utility of a brief online educational intervention for promoting adolescent mental health during important life transitions.

One important factor that appears to be associated with wellbeing and resilience is that of beliefs about growth and response to failure. Individuals often respond to challenge by either a) retreating and/or making negative attributions about themselves or others, or b) view challenge as an opportunity for learning and growth, and not consider failure to be an indication of personal shortcomings. The difference between these two responses to challenge reflects beliefs about the malleability of personal characteristics; these beliefs are referred to as "implicit theories" or more colloquially "mindset". Those who hold "entity" theories (fixed mindset) believe personal characteristics are stable and unchanging, while those with a malleable or "incremental theories" (growth mindset) believe personal characteristics are changeable and can be developed through effort and learning . Research has broadly suggested that those with entity theories may be more prone to experience difficulties and be at risk for mental illness, while those with incremental theories experience greater resilience and well-being.

Previous research has indicated that incremental theory can be taught via educational interventions, and increasing belief in incremental theory has been associated with positive effects. Further, integrating positive psychology into educational institutions to foster youth development has been recommended by many researchers. Youth spend substantial amounts of time in school, making schools an appropriate setting for interventions that aim to promote well-being and prevent mental illness. Thus, this study will test the effects of a brief implicit theory intervention on well-being and depressive symptoms.The intervention is similar to previous implicit theory interventions and teaches youth an incremental theory of socially relevant characteristics (i.e., that people can change and that personal attributes are malleable).

Implicit theory of personality (ie, beliefs about the malleability of personal attributes and socially relevant characteristics) has also been associated with depressive symptoms in youth. In a study of grade 9 students, researchers found that a brief intervention that taught incremental theory of personality (that personal attributes can grow and change) was associated with stability of reported levels of depressive symptoms over 9 months. In this intervention, students read a compelling article that demonstrated incremental theory of either personality (experimental) or athletic ability (control), then students were asked to summarize the lesson of the article and apply their own experience. Over time (9 months) those in the control condition showed an increase in depressive symptoms while those exposed to the incremental theory of personality did not show the same increase, and incidence of clinically significant depressive symptoms remained stable. The increase seen in the control group was noted to be proportional to that commonly experienced by those transitioning to high school, suggesting the intervention may have promise for successfully ameliorating developmentally typical increases in depressive symptoms. Although this brief intervention was associated with significant positive outcomes, replication and application to other samples at risk for depressive symptoms (such as youth transitioning out of high school and to post secondary education) is warranted. Towards this end, the current study will examine the impact of an intervention that teaches incremental theory on well-being and depressive symptoms in students in the first and last years of high school.

ELIGIBILITY:
Inclusion Criteria:

* A student at one of the recruited schools in grade 9 or 12
* Age 13-18 years
* Able to read and write fluently in English
* Have parent/guardian consent, and provide participant consent

Exclusion Criteria:

* Not a registered student at one of the recruited schools
* Less than 13 or more than 18 years old
* Unable to read and write fluently in English
* Does not have parent/guardian consent or does not consent to participate

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 576 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | 4 months (Oct 2019 - Feb 2020)
  Score on the Beck Depression Inventory-II. The BDI-II consists of 21 items using a 4-point Likert scale from 0 to 3, however the current study will use only 19 items. The item querying suicidal ideation will be removed, as this may be triggering, and researchers would not be able to follow up with those who would highly endorse this item. The item querying sexual interest will be removed, as this may not be equally applicable across the sample. Scores on each item are summed to determine summary scores from 0-57. Higher scores indicate higher levels of depressive symptoms.
Perceived happiness | 4 months (Oct 2019 - Feb 2020)
  score on the Subjective Happiness Scale (SHS). This measure consists of four items measured on a 7-point Likert scale; responses are averaged to create a summary score (minimum=1, maximum=7) and higher scores reflect higher levels of subjective happiness.
Life satisfaction | 4 months (Oct 2019 - Feb 2020)
  score on the Brief Multidimensional Student Life Satisfaction Scale (BMSLSS). The BMSLSS includes five items that assess global life satisfaction as a reflection of five life domains: family, school, friends, self, and living environment. The BMSLSS uses a 7-point Likert scale that ranges from delighted to terrible. The score of each item will be averaged to create a single score (minimum=1, maximum=7) such that higher scores represent higher levels of life satisfaction.

SECONDARY OUTCOMES:
Implicit theory of personality | immediately post administration of the intervention
  Score on the Implicit Personality Theory Questionnaire. This is a three-item measure that uses a 6-point Likert scale that ranges from strongly agree to strongly disagree to measure the extent individuals believe one's personality can change. The score of each item will be averaged to create a single score (minimum=1, maximum=6) such that higher values will be associated with higher levels of entity beliefs.
Implicit theory of a person (general) | Immediately post administration of the intervention
  Score on the Implicit Person Measure. This is a three item measure with a 6-point Likert scale ranging from strongly agree to strongly disagree. Scores on each item will be averaged to create a single score (minimum=1, maximum=6), and higher average scores will be associated with more entity beliefs.
Implicit theory of personality | 4 months (Oct 2019 - Feb 2020)
  Score on the Implicit Personality Theory Questionnaire. This is a three-item measure that uses a 6-point Likert scale that ranges from strongly agree to strongly disagree to measure the extent individuals believe one's personality can change. The score of each item will be averaged to create a single score (minimum=1, maximum=6) such that higher values will be associated with higher levels of entity beliefs.
Implicit theory of a person (general) | 4 months (Oct 2019 - Feb 2020)
  Score on the Implicit Person Measure. This is a three item measure with a 6-point Likert scale ranging from strongly agree to strongly disagree. Scores on each item will be averaged to create a single score (minimum=1, maximum=6), and higher average scores will be associated with more entity beliefs.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Lumley, PhD, Principal Investigator — University of Guelph
Locations (1):
- University of Guelph, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data as this has not been approved by our Research Ethics Board

REFERENCES:
- [Background] Abela, J. R. Z., & Hankin, B. L. (2008). Depression in children and adolescents: Causes, treatment, and prevention. In J. R. Z. Abela & B. L. Hankin (Eds.), Handbook of depression in children and adolescents (pp. 3-5). New York, NY, US: The Guilford Press.
- [Background] Abramson, L. Y., Metalsky, G. I., & Alloy, L. B. (1989). Hopelessness depression: A theory-based subtype of depression. Psychological review, 96(2), 358.
- [Background] Abramson LY, Seligman ME, Teasdale JD. Learned helplessness in humans: critique and reformulation. J Abnorm Psychol. 1978 Feb;87(1):49-74. No abstract available. PMID 649856
- [Background] Dweck, C. S., Chiu, C. Y., & Hong, Y. Y. (1995). Implicit theories and their role in judgments and reactions: A word from two perspectives. Psychological inquiry, 6(4), 267-285.
- [Background] Dweck, C. S., & Leggett, E. L. (1988). A social-cognitive approach to motivation and personality. Psychological review, 95(2), 256.
- [Background] Furlong, M. J., Gilman, R., & Huebner, E. S. (2014). Handbook of Positive Psychology in Schools, 2nd Ed New York. NY: Taylor & Francis.
- [Background] Greenberg MT, Weissberg RP, O'Brien MU, Zins JE, Fredericks L, Resnik H, Elias MJ. Enhancing school-based prevention and youth development through coordinated social, emotional, and academic learning. Am Psychol. 2003 Jun-Jul;58(6-7):466-74. doi: 10.1037/0003-066x.58.6-7.466. PMID 12971193
- [Background] Hankin BL, Abramson LY, Moffitt TE, Silva PA, McGee R, Angell KE. Development of depression from preadolescence to young adulthood: emerging gender differences in a 10-year longitudinal study. J Abnorm Psychol. 1998 Feb;107(1):128-40. doi: 10.1037//0021-843x.107.1.128. PMID 9505045
- [Background] Hong, Y. Y., Chiu, C. Y., Dweck, C. S., Lin, D. M. S., & Wan, W. (1999). Implicit theories, attributions, and coping: A meaning system approach. Journal of Personality and Social psychology, 77(3), 588.
- [Background] Masten, A., Herbers, J., Cutuli, J., & Lafavor, T. (2008). Promoting competence and resilience in the school context. Professional School Counseling, 12(2), 76-84.
- [Background] Merikangas KR, He JP, Burstein M, Swanson SA, Avenevoli S, Cui L, Benjet C, Georgiades K, Swendsen J. Lifetime prevalence of mental disorders in U.S. adolescents: results from the National Comorbidity Survey Replication--Adolescent Supplement (NCS-A). J Am Acad Child Adolesc Psychiatry. 2010 Oct;49(10):980-9. doi: 10.1016/j.jaac.2010.05.017. Epub 2010 Jul 31. PMID 20855043
- [Background] Petersen AC, Compas BE, Brooks-Gunn J, Stemmler M, Ey S, Grant KE. Depression in adolescence. Am Psychol. 1993 Feb;48(2):155-68. doi: 10.1037//0003-066x.48.2.155. PMID 8442570
- [Background] Rindfuss RR. The young adult years: diversity, structural change, and fertility. Demography. 1991 Nov;28(4):493-512. No abstract available. PMID 1769399
- [Background] Seligman, M. E., Ernst, R. M., Gillham, J., Reivich, K., & Linkins, M. (2009). Positive education: Positive psychology and classroom interventions. Oxford review of education, 35(3), 293-311.
- [Background] Yeager, D. S., & Dweck, C. S. (2012). Mindsets that promote resilience: When students believe that personal characteristics can be developed. Educational psychologist, 47(4), 302-314.
- [Result] Blackwell LS, Trzesniewski KH, Dweck CS. Implicit theories of intelligence predict achievement across an adolescent transition: a longitudinal study and an intervention. Child Dev. 2007 Jan-Feb;78(1):246-63. doi: 10.1111/j.1467-8624.2007.00995.x. PMID 17328703
- [Result] Burnette JL, Russell MV, Hoyt CL, Orvidas K, Widman L. An online growth mindset intervention in a sample of rural adolescent girls. Br J Educ Psychol. 2018 Sep;88(3):428-445. doi: 10.1111/bjep.12192. Epub 2017 Sep 27. PMID 28960257
- [Result] Miu, A. S., & Yeager, D. S. (2015). Preventing symptoms of depression by teaching adolescents that people can change: Effects of a brief incremental theory of personality intervention at 9-month follow-up. Clinical Psychological Science, 3(5), 726-743.